CLINICAL TRIAL: NCT05134194
Title: A Muti-center, Open-label, Randomized, Phase III Study of Camrelizumab Plus Treatment of Physician Choice Versus Treatment of Physician Choice for Metastatic Triple-Negative Breast Cancer Who Received at Least Two Prior Systemic Chemotherapy Regimens for Advanced/Metastatic Setting
Brief Title: A Study of Camrelizumab in Combination With Chemotherapy Regimen Comparative Chemotherapy Regimen for Metastatic Triple-negative Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment]
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-327
Record Dates: First submitted 2021-11-09; First posted 2021-11-24 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to Arm A (Camrelizumab+Capecitabine or Eribulin or Gemcitabine or Vinorelbine), Arm B (Capecitabine or Eribulin or Gemcitabine or Vinorelbine)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Camrelizumab in combination with capecitabine or eribulin or gemcitabine or vinorelbine
  Interventions: Drug: Camrelizumab、Capecitabine/eribulin/gemcitabine/vinorelbine
- Arm B (Experimental): Capecitabine or eribulin or gemcitabine or vinorelbine
  Interventions: Drug: Capecitabine/eribulin/gemcitabine/vinorelbine

INTERVENTIONS:
Drug: Camrelizumab、Capecitabine/eribulin/gemcitabine/vinorelbine — Camrelizumab in combination with capecitabine or eribulin or gemcitabine or vinorelbine
  Arms: Arm A
Drug: Capecitabine/eribulin/gemcitabine/vinorelbine — Capecitabine or eribulin or gemcitabine or vinorelbine
  Arms: Arm B

SUMMARY:
Approximately 104 subjects with recurrent or metastatic IM triple negative breast cancer were planned to be included in the study, and screened eligible subjects were randomly assigned in a 1:1 ratio to treatment with the combination of Camrelizumab and investigator's choice of chemotherapy (test arm), treatment with investigator's choice of chemotherapy (control arm), and the stratification factor was liver metastasis (with vs without). After enrollment, subjects in the test group were treated with Camrelizumab 200 mg IV every 3 weeks for one cycle. The investigator's choice of single agent chemotherapy regimen (capecitabine, eribulin, gemcitabine, or vinorelbine) was every 3 weeks for one cycle until disease progression, intolerable toxicity, withdrawal of informed consent, or discontinuation at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG Performance Status of 0-1.
2. Expected lifetime of not less than three months
3. Metastatic triple negative invasive breast cancer, confirmed by histopathological testing, was diagnosed as triple negative according to the American Society of Clinical Oncology / College of American Pathologists (ASCO / CAP) guidelines for pathological typing.
4. Target lesions with at least one measurable diameter line were present as judged by the investigator on imaging (RECIST v1.1 criteria).
5. The major organs function well.
6. Women of childbearing age were required to have a serum pregnancy study within 7 days prior to first dose and be assessed as nonpregnant. Women of reproductive age subjects were required to agree to a highly effective method of contraception during the study and for 6 months after the last administration of study drug.
7. Volunteered to join this study, signed informed consent, had good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

1. Known central nervous system (CNS) disease.
2. Uncontrollable moderate to large amounts of pleural effusion requiring repeated drainage, peritoneal effusion, or pericardial effusion.
3. Any subject with known or suspected autoimmune disease other than: hypothyroidism due to autoimmune thyroiditis requiring hormone replacement therapy only; Subjects with stable type I diabetes in whom glycemia was controlled.
4. Within 6 months prior to randomization, the following conditions occurred: myocardial infarction, severe / unstable angina, cardiac insufficiency of NYHA class 2 and above, clinically significant supraventricular or ventricular arrhythmia requiring intervention, and symptomatic congestive heart failure.
5. Previous or current history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, idiopathic interstitial pneumonia, or evidence of active pneumonia on chest CT screening; Patients with a history of radiation pneumonitis (fibrosis) in the irradiated field were excluded.
6. History of live attenuated influenza vaccination within 28 days before first dose of study medication or anticipated during the study.
7. Human immunodeficiency virus (HIV) infection or known to have acquired immune deficiency syndrome (AIDS); Active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU / ml; hepatitis C, defined as HCV-RNA above the lower limit of detection of the analytical method) or coinfection with hepatitis B and C.
8. Presence of severe infection including, but not limited to, bacteremia requiring hospitalization, severe pneumonia within 4 weeks prior to first dose; With evidence of active tuberculosis infection within 1 year before drug administration.
9. Had a diagnosis of any other malignancy within 5 years before study entry, with the exception of adequately treated basal cell carcinoma or squamous cell skin carcinoma, or carcinoma in situ of the cervix.
10. Major surgery within 28 days before randomization (tissue biopsy required for diagnosis and placement of a central venous catheter operation [PICC] via peripheral venipuncture were permitted).
11. Patients who had previously received or were ready to undergo allogeneic bone marrow transplantation or solid organ transplantation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Treatment was assessed every 6 weeks after treatment initiation（up to 30 weeks）, regardless of whether treatment was delayed or interrupted, until disease progression or study end, whichever occurred first.
  assessed by independent imaging (IRC), according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided